CLINICAL TRIAL: NCT06585436
Title: Selective Versus Stepwise Removal of Deep Carious Lesions in Permanent Teeth Using Different Medicaments: An in Vivo Study
Brief Title: Selective Versus Stepwise Removal of Deep Carious Lesions in Permanent Teeth Using Different Medicaments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Abdallah Rabiea, teaching assistant, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2/9/2022
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Caries Arrested

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- selective removal (chitosan loaded nano hydroxyapatite ) (Experimental): selective removal then apply chitosan loaded nano hydroxyapatite
  Interventions: Procedure: partial caries removal
- selective removal (nano bioactive glass/GIC) (Experimental): selective removal then apply (nano bioactive glass/GIC)
  Interventions: Procedure: partial caries removal
- selective removal (nanosilver) (Experimental): selective removal then apply (nanosilver)
  Interventions: Procedure: partial caries removal
- stepwise removal (chitosan loaded nano hydroxyapatite ) (Experimental): stepwise removal then apply (chitosan loaded nano hydroxyapatite )
  Interventions: Procedure: partial caries removal
- stepwise removal (nano bioactive glass/GIC) (Experimental): selective removal (nano bioactive glass/GIC)
  Interventions: Procedure: partial caries removal
- stepwise removal (nanosilver) (Experimental): selective removal then apply (nanosilver)
  Interventions: Procedure: partial caries removal

INTERVENTIONS:
Procedure: partial caries removal — removal of all cavity caries except last layer related to the pulp

SUMMARY:
The study involved 54 adult patients between the ages of 18 and 50 years who had a posterior permanent tooth with a deep occlusal (Class I) carious lesion that extended to the inner third of the dentin (D3) and divided them into two equal groups randomly (N=27) according to the caries removal technique: group 1 (SE), and group 2 (SW). Then each main group was equally subdivided into three equal subgroups (n=9) according to the applied dentin dressing material as follows: Subgroup 1: Nano-silver compound (NSC), Subgroup 2: Chitosan-loaded nano hydroxy apatite (CS/N-HAp), Subgroup 3: Bioactive glass ionomer (N-BAG/GIC). At the first visit both groups received the same treatment of incomplete caries excavation, application of dentin dressing materials and sealing temporarily for 3-months with a glass ionomer cement (GIC). At the second visit the GIC reduced pulpally in (SE) group leaving 2 mm as base and completely removal the remaining carious lesion in (SW) group then re-application of same dentin dressing material on each tooth and GIC as a base. Finally, all cavities were restored with selective enamel etching technique, after which self-etch adhesive and Nano-filled composite resin are applied according to manufacturer instructions. The clinical and digital radiographic evaluations of the success and failure rates were performed at: baseline (7 days), 3, 12, and 18-months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with first and second molars with occlusal deep carious lesions (Class I) extending to the inner third of dentin thickness on radiographic examination using (i-sensor H1, Woodpecker, China).
2. Teeth with a healthy response to the electrical pulp tester (DY 310, Denjoy Dental CO., LTD, China).
3. Teeth with the absence of spontaneous pain.
4. Teeth with a negative sensitivity to percussion.
5. Teeth with the absence of periapical lesions by a digital radiographic examination.
6. Clinically, all teeth were without any mobility.
7. Patients who will complete the procedure of follow up.
8. Patients who will sign the consent.

Exclusion Criteria:

1. Mutilated teeth or teeth with caries extending subgingivally.
2. Teeth with the existence of previous restorations.
3. Teeth with periodontal disease, any swelling, fistulas, signs of irreversible pulpitis or necrotic pulp.
4. Teeth with roots showing external or internal resorption.
5. Pregnant women.
6. Presence of any systemic disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
post operative pain | 7 days
  evaluation of the post operative pain following restorations using modified USPHS
post operative pain | 3 months
  evaluation of the post operative pain following restorations using modified USPHS
post operative pain | 12 months
  evaluation of the post operative pain following restorations using modified USPHS
post operative pain | 18 months
  evaluation of the post operative pain following restorations using modified USPHS

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar university, Cairo, Egypt